CLINICAL TRIAL: NCT01559467
Title: The Supplementary Role of Cardiovascular Magnetic Resonance Imaging and Computed Tomography Angiography to Routine Clinical Practice in Suspected Non-ST Elevation Myocardial Infarction - A Randomized Controlled Trial
Brief Title: The Supplementary Role of Non-invasive Imaging to Routine Clinical Practice in Suspected Non-ST-elevation Myocardial Infarction
Acronym: CARMENTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Dutch Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL37574.068.11 / METC 11-2-077
Record Dates: First submitted 2012-03-12; First posted 2012-03-21 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2016-07

CONDITIONS: Chest Pain; Myocardial Infarction; Acute Coronary Syndrome; Coronary Artery Disease; Myocardial Ischemia
Keywords: Myocardial infarction; Randomized Controlled Trial; Magnetic Resonance Imaging; Coronary Angiography; Tomography, X-Ray Computed; Mortality; Complications; Quality of Life; Cost-Benefit Analysis
MeSH Terms: conditions — Chest Pain; Myocardial Infarction; Acute Coronary Syndrome; Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Routine clinical care plus early CMR (Other)
  Interventions: Other: Cardiovascular Magnetic Resonance Imaging
- Routine clinical care (No Intervention)
- Routine clinical care plus early CTA (Other)
  Interventions: Other: Computed Tomography Angiography

INTERVENTIONS:
Other: Cardiovascular Magnetic Resonance Imaging — Routine clinical care plus cardiovascular magnetic resonance imaging early in the diagnostic process
  Arms: Routine clinical care plus early CMR
Other: Computed Tomography Angiography — Routine clinical care plus computed tomography angiography early in the diagnostic process
  Arms: Routine clinical care plus early CTA

SUMMARY:
Approximately half of patients with acute chest pain, a very common reason for emergency department visits worldwide, have a cardiac cause. Two-thirds of patients with a cardiac cause are eventually diagnosed with a so-called non-ST-elevation myocardial infarction. The diagnosis of non-ST-elevation myocardial infarction is based on a combination of symptoms, electrocardiographic changes, and increased serum cardiac specific biomarkers (high-sensitive troponin T). Although being very sensitive of myocardial injury, increased high-sensitive troponin T levels are not specific for myocardial infarction. Invasive coronary angiography is still the reference standard for coronary imaging in suspected non-ST-elevation myocardial infarction. This study investigates whether non-invasive imaging early in the diagnostic process (computed tomography angiography (CTA) or cardiovascular magnetic resonance imaging (CMR)) can prevent unnecessary invasive coronary angiography. For this, patients will be randomly assigned to either one of three strategies: 1) routine clinical care and computed tomography angiography early in the diagnostic process, 2) routine clinical care and cardiovascular magnetic resonance imaging early in the diagnostic process, or 3) routine clinical care without non-invasive imaging early in the diagnostic process.

ELIGIBILITY:
Inclusion Criteria:

* Prolonged symptoms suspected of cardiac origin (angina pectoris or angina equivalent), and presentation on the cardiac emergency department <24 hours after symptom onset

  * Increased levels of high-sensitive Troponin-T (>14ng/L)
  * Age >18 years and <85 years
  * Willing and capable to give written informed consent
  * Written informed consent

Exclusion Criteria:

* Ongoing severe ischemia requiring immediate invasive coronary angiography
* Shock (mean arterial pressure < 60 mmHg) or severe heart failure (Killip Class ≥ III)
* ST-elevation myocardial infarction (ST-elevation in 2 contiguous leads: ≥0.2mV in men or ≥0.15 mV in women in leads V2-V3 and/or ≥0.1 mV in other leads or new left bundle branch block)
* Chest pain highly suggestive of non-cardiac origin:

  * Acute aortic dissection
  * Acute pulmonary embolism (high risk patient defined as Wells score >6)
  * Musculoskeletal or gastro-intestinal pain
  * Other (pneumothorax, pneumonia, rib fracture, etc.)
* Previously known coronary artery disease, defined as:

  * Any non-invasive diagnostic imaging test positive for coronary artery disease
  * Coronary stenosis >50% on any previous invasive coronary angiography or computed tomography angiography
  * Documented previous myocardial infarction
  * Documented previous coronary artery revascularization
  * Known cardiomyopathy
* Pregnancy
* Life threatening arrhythmia on the cardiac emergency department or prior to presentation
* Tachycardia (≥100/bpm)
* Atrial fibrillation
* Angina pectoris secondary to anemia (<5.6 mmol/L), untreated hyperthyroidism, aortic valve stenosis (aortic valve area ≤ 1.5 cm2), or severe hypertension (>200/110 mmHg)
* Life expectancy <1 year (malignancy, etc.)
* Contraindications to cardiovascular magnetic resonance imaging: metallic implant (vascular clip, neuro-stimulator, cochlear implant), pacemaker or implantable cardiac defibrillator, claustrophobia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-04; Primary Completion 2017-05 (Actual); Study Completion 2017-06-19 (Actual)

PRIMARY OUTCOMES:
Total number of patients with at least one invasive coronary angiography during initial admission | During initial hospital admission, an expected average of 7 days

SECONDARY OUTCOMES:
Thirty-day clinical outcome (a composite of major adverse cardiac events [MACE] and major procedure related complications) | 30 days
One-year clinical outcome (a composite of major adverse cardiac events [MACE] and major procedure related complications) | One-year
Quality of life | One-year
Cost-effectiveness | After study completion, expected after 3 years
  The economic evaluation will be a cost-effectiveness analysis, with quality-adjusted life years (QALYs) as outcome measure. Effects will be calculated in terms of QALYs. To investigate the cost-effectiveness of the three strategies, incremental cost-effectiveness ratios (ICERs) will be calculated. Cost-effectiveness acceptability curves (CEACs) are derived in order to show the probability of each strategy being the optimal choice, for a range of possible maximum values a decision maker is willing to pay for a QALY.
Cardiogoniometry | After study completion, expected after 3 years
  A retrospective analysis will be performed to investigate whether CGM performed on the cardiac emergency department can differentiate between a coronary and non-coronary etiology in suspected NSTEMI

CONTACTS AND LOCATIONS:
Overall Officials: Harry J Crijns, MD, PhD, Principal Investigator — Maastricht University Medical Center; Joachim Wildberger, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Hamm CW, Goldmann BU, Heeschen C, Kreymann G, Berger J, Meinertz T. Emergency room triage of patients with acute chest pain by means of rapid testing for cardiac troponin T or troponin I. N Engl J Med. 1997 Dec 4;337(23):1648-53. doi: 10.1056/NEJM199712043372302. PMID 9385123
- [Background] Reichlin T, Hochholzer W, Bassetti S, Steuer S, Stelzig C, Hartwiger S, Biedert S, Schaub N, Buerge C, Potocki M, Noveanu M, Breidthardt T, Twerenbold R, Winkler K, Bingisser R, Mueller C. Early diagnosis of myocardial infarction with sensitive cardiac troponin assays. N Engl J Med. 2009 Aug 27;361(9):858-67. doi: 10.1056/NEJMoa0900428. PMID 19710484
- [Background] Kim HW, Farzaneh-Far A, Kim RJ. Cardiovascular magnetic resonance in patients with myocardial infarction: current and emerging applications. J Am Coll Cardiol. 2009 Dec 29;55(1):1-16. doi: 10.1016/j.jacc.2009.06.059. PMID 20117357
- [Background] Anderson JL, Adams CD, Antman EM, Bridges CR, Califf RM, Casey DE Jr, Chavey WE 2nd, Fesmire FM, Hochman JS, Levin TN, Lincoff AM, Peterson ED, Theroux P, Wenger NK, Wright RS, Smith SC Jr; 2011 WRITING GROUP MEMBERS; ACCF/AHA TASK FORCE MEMBERS. 2011 ACCF/AHA Focused Update Incorporated Into the ACC/AHA 2007 Guidelines for the Management of Patients With Unstable Angina/Non-ST-Elevation Myocardial Infarction: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. Circulation. 2011 May 10;123(18):e426-579. doi: 10.1161/CIR.0b013e318212bb8b. Epub 2011 Mar 28. No abstract available. PMID 21444888
- [Background] Hoenig MR, Aroney CN, Scott IA. Early invasive versus conservative strategies for unstable angina and non-ST elevation myocardial infarction in the stent era. Cochrane Database Syst Rev. 2010 Mar 17;(3):CD004815. doi: 10.1002/14651858.CD004815.pub3. PMID 20238333
- [Background] Ricciardi MJ, Wu E, Davidson CJ, Choi KM, Klocke FJ, Bonow RO, Judd RM, Kim RJ. Visualization of discrete microinfarction after percutaneous coronary intervention associated with mild creatine kinase-MB elevation. Circulation. 2001 Jun 12;103(23):2780-3. doi: 10.1161/hc2301.092121. PMID 11401931
- [Background] Kwong RY, Schussheim AE, Rekhraj S, Aletras AH, Geller N, Davis J, Christian TF, Balaban RS, Arai AE. Detecting acute coronary syndrome in the emergency department with cardiac magnetic resonance imaging. Circulation. 2003 Feb 4;107(4):531-7. doi: 10.1161/01.cir.0000047527.11221.29. PMID 12566362
- [Background] Leurent G, Langella B, Fougerou C, Lentz PA, Larralde A, Bedossa M, Boulmier D, Le Breton H. Diagnostic contributions of cardiac magnetic resonance imaging in patients presenting with elevated troponin, acute chest pain syndrome and unobstructed coronary arteries. Arch Cardiovasc Dis. 2011 Mar;104(3):161-70. doi: 10.1016/j.acvd.2011.01.005. Epub 2011 Apr 2. PMID 21497305
- [Background] Meijboom WB, Mollet NR, Van Mieghem CA, Weustink AC, Pugliese F, van Pelt N, Cademartiri F, Vourvouri E, de Jaegere P, Krestin GP, de Feyter PJ. 64-Slice CT coronary angiography in patients with non-ST elevation acute coronary syndrome. Heart. 2007 Nov;93(11):1386-92. doi: 10.1136/hrt.2006.112771. Epub 2007 Mar 7. PMID 17344332
- [Background] Vanhoenacker PK, Decramer I, Bladt O, Sarno G, Bevernage C, Wijns W. Detection of non-ST-elevation myocardial infarction and unstable angina in the acute setting: meta-analysis of diagnostic performance of multi-detector computed tomographic angiography. BMC Cardiovasc Disord. 2007 Dec 19;7:39. doi: 10.1186/1471-2261-7-39. PMID 18093295
- [Background] Hoffmann U, Bamberg F, Chae CU, Nichols JH, Rogers IS, Seneviratne SK, Truong QA, Cury RC, Abbara S, Shapiro MD, Moloo J, Butler J, Ferencik M, Lee H, Jang IK, Parry BA, Brown DF, Udelson JE, Achenbach S, Brady TJ, Nagurney JT. Coronary computed tomography angiography for early triage of patients with acute chest pain: the ROMICAT (Rule Out Myocardial Infarction using Computer Assisted Tomography) trial. J Am Coll Cardiol. 2009 May 5;53(18):1642-50. doi: 10.1016/j.jacc.2009.01.052. PMID 19406338
- [Derived] van Cauteren YJM, Smulders MW, Theunissen RALJ, Gerretsen SC, Adriaans BP, Bijvoet GP, Mingels AMA, van Kuijk SMJ, Schalla S, Crijns HJGM, Kim RJ, Wildberger JE, Heijman J, Bekkers SCAM. Cardiovascular magnetic resonance accurately detects obstructive coronary artery disease in suspected non-ST elevation myocardial infarction: a sub-analysis of the CARMENTA Trial. J Cardiovasc Magn Reson. 2021 Mar 22;23(1):40. doi: 10.1186/s12968-021-00723-6. PMID 33752696
- [Derived] Smulders MW, Kietselaer BLJH, Wildberger JE, Dagnelie PC, Brunner-La Rocca HP, Mingels AMA, van Cauteren YJM, Theunissen RALJ, Post MJ, Schalla S, van Kuijk SMJ, Das M, Kim RJ, Crijns HJGM, Bekkers SCAM. Initial Imaging-Guided Strategy Versus Routine Care in Patients With Non-ST-Segment Elevation Myocardial Infarction. J Am Coll Cardiol. 2019 Nov 19;74(20):2466-2477. doi: 10.1016/j.jacc.2019.09.027. PMID 31727284
- [Derived] Smulders MW, Kietselaer BL, Das M, Wildberger JE, Crijns HJ, Veenstra LF, Brunner-La Rocca HP, van Dieijen-Visser MP, Mingels AM, Dagnelie PC, Post MJ, Gorgels AP, van Asselt AD, Vogel G, Schalla S, Kim RJ, Bekkers SC. The role of cardiovascular magnetic resonance imaging and computed tomography angiography in suspected non-ST-elevation myocardial infarction patients: design and rationale of the CARdiovascular Magnetic rEsoNance imaging and computed Tomography Angiography (CARMENTA) trial. Am Heart J. 2013 Dec;166(6):968-75. doi: 10.1016/j.ahj.2013.09.012. Epub 2013 Oct 23. PMID 24268210